CLINICAL TRIAL: NCT01059825
Title: A 12-Week, Phase 2, Randomized, Double-Blinded, Placebo-Controlled, Dose-Ranging, Parallel Group Study to Evaluate the Safety, Tolerability and Efficacy Of Once Daily PF-04971729 And Sitagliptin On Glycemic Control And Body Weight In Adult Patients With Type 2 Diabetes Mellitus Inadequately Controlled On Metformin
Brief Title: Study Of Safety And Efficacy Of Ertugliflozin (PF-04971729, MK-8835) In Participants With Type 2 Diabetes (MK-8835-016)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-016; B1521006 (Other: Pfizer protocol number); 2009-017131-18 (EudraCT Number)
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Phase 2; safety and efficacy study with ertugliflozin (PF-04971729, MK-8835); Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Placebo for ertugliflozin (1 mg or 5 mg and 25 mg) and placebo to sitagliptin, oral, once daily for 84 days
  Interventions: Drug: Placebo to Ertugliflozin; Drug: Placebo to Sitagliptin; Drug: Metformin
- Ertugliflozin 1 mg (Experimental): Ertugliflozin 1 mg, placebo for ertugliflozin (1 mg or 5 mg and 25 mg), and placebo to sitagliptin, oral, once daily for 84 days
  Interventions: Drug: Placebo to Ertugliflozin; Drug: Ertugliflozin 1 mg; Drug: Placebo to Sitagliptin; Drug: Metformin
- Ertugliflozin 5 mg (Experimental): Ertugliflozin 5 mg, placebo for ertugliflozin (1 mg or 5 mg and 25 mg), and placebo to sitagliptin, oral, once daily for 84 days
  Interventions: Drug: Placebo to Ertugliflozin; Drug: Ertugliflozin 5 mg; Drug: Placebo to Sitagliptin; Drug: Metformin
- Ertugliflozin 10 mg (Experimental): Ertugliflozin 10 mg, placebo for ertugliflozin (25 mg), and placebo to sitagliptin, oral, once daily for 84 days
  Interventions: Drug: Placebo to Ertugliflozin; Drug: Ertugliflozin 5 mg; Drug: Placebo to Sitagliptin; Drug: Metformin
- Ertugliflozin 25 mg (Experimental): Ertugliflozin 25 mg, placebo for ertugliflozin (1 mg or 5 mg), and placebo to sitagliptin, oral, once daily for 84 days
  Interventions: Drug: Placebo to Ertugliflozin; Drug: Ertugliflozin 25 mg; Drug: Placebo to Sitagliptin; Drug: Metformin
- Sitagliptin 100 mg (Active Comparator): Sitagliptin 100 mg, placebo for ertugliflozin (1 mg or 5 mg and 25 mg), oral, once daily for 84 days
  Interventions: Drug: Placebo to Ertugliflozin; Drug: Sitagliptin 100 mg; Drug: Metformin

INTERVENTIONS:
Drug: Placebo to Ertugliflozin — Tablet(s), 1 or 2, matching placebo to 1-mg, 5-mg and/or 25-mg tablets, once daily for 84 days
Drug: Ertugliflozin 1 mg — Tablet, 1 mg, once daily for 84 days
  Arms: Ertugliflozin 1 mg
Drug: Ertugliflozin 5 mg — Tablet(s), 1 or 2, 5-mg tablets once daily for 84 days
  Arms: Ertugliflozin 10 mg; Ertugliflozin 5 mg
Drug: Ertugliflozin 25 mg — Tablet, 25 mg, once daily for 84 days
  Arms: Ertugliflozin 25 mg
Drug: Sitagliptin 100 mg — Tablet, 100 mg, once daily for 84 days
  Other Names: Januvia®, Tesavel®, Xelevia®, Ristaben®
  Arms: Sitagliptin 100 mg
Drug: Placebo to Sitagliptin — Tablet, matching placebo to 100 mg, once daily for 84 days
  Arms: Ertugliflozin 1 mg; Ertugliflozin 10 mg; Ertugliflozin 25 mg; Ertugliflozin 5 mg; Placebo
Drug: Metformin — Participants continued pre-study stable doses of metformin during the run-in and treatment periods of the study (maximum dose up to 2500 mg/day or 3000 mg/day where the maximum metformin dose per the local country product labels was 3000 mg/day).
  Other Names: Fortamet®, Glucophage®, Glucophage® XR, Glumetza®, Riomet®, Metgluco®, Glycoran®

SUMMARY:
MK-8835-016 (B1521006) is designed to evaluate the safety and efficacy of an investigational drug, ertugliflozin (MK-8835, PF-04971729) in participants with Type 2 diabetes mellitus. Participants in the study will receive 1 of 6 treatments for 12 weeks including 1 treatment with an approved drug (sitagliptin) for the treatment of Type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Participants with type 2 diabetes on stable doses of background medicines for management of the diabetes; aged 18-70 years; body mass index between 23-45 kg/m^2

Exclusion Criteria:

* Participants with type 1 diabetes, heart attack or stroke in last 6-months, uncontrolled blood pressure, significant kidney disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2010-02-24 (Actual); Primary Completion 2011-01-20 (Actual); Study Completion 2011-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Amin NB, Wang X, Jain SM, Lee DS, Nucci G, Rusnak JM. Dose-ranging efficacy and safety study of ertugliflozin, a sodium-glucose co-transporter 2 inhibitor, in patients with type 2 diabetes on a background of metformin. Diabetes Obes Metab. 2015 Jun;17(6):591-598. doi: 10.1111/dom.12460. Epub 2015 Mar 31. PMID 25754396
- [Derived] Fediuk DJ, Sahasrabudhe V, Dawra VK, Zhou S, Sweeney K. Population Pharmacokinetic Analyses of Ertugliflozin in Select Ethnic Populations. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1297-1306. doi: 10.1002/cpdd.970. Epub 2021 Jul 2. PMID 34213819

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 375 enrolled participants included in the metformin run-in period, 328 participants were randomized to 1 of 6 treatment groups.
Groups:
- Metformin Run-in: Participants received open-label metformin during the run-in period.
Period: Enrolled, Run-in Period
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg | Metformin Run-in
Started | 0 | 0 | 0 | 0 | 0 | 0 | 375
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 328
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 47
Not completed — Adverse event not related to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Did not meet entrance criteria | 0 | 0 | 0 | 0 | 0 | 0 | 14
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 13
Not completed — Other reason not specified | 0 | 0 | 0 | 0 | 0 | 0 | 7
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 5
Period: Treatment Period
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg | Metformin Run-in
Started | 54 (54 participants who completed the run-in period were randomized to this treatment group.) | 54 (54 participants who completed the run-in period were randomized to this treatment group.) | 55 (55 participants who completed the run-in period were randomized to this treatment group.) | 55 (55 participants who completed the run-in period were randomized to this treatment group.) | 55 (55 participants who completed the run-in period were randomized to this treatment group.) | 55 (55 participants who completed the run-in period were randomized to this treatment group.) | 0 (Participants who completed run-in were randomized to 1 of 6 treatment groups.)
Completed | 44 | 50 | 49 | 44 | 47 | 52 | 0
Not Completed | 10 | 4 | 6 | 11 | 8 | 3 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 5 | 4 | 1 | 0
Not completed — Other reason not specified | 1 | 2 | 1 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 1 | 1 | 0
Not completed — Adverse event related to study drug | 1 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Insufficient clinical response | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse event not related to study drug | 0 | 1 | 2 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Of the 375 enrolled participants included in the metformin run-in period, 328 participants were randomized to 1 of 6 treatment groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg | Total
Number analyzed (Participants) | 54 | 54 | 55 | 55 | 55 | 55 | 328
Age, Customized [Number; unit: Participants]
  < 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-44 years | 8 | 10 | 6 | 1 | 9 | 13 | 47
  45-64 years | 41 | 36 | 42 | 47 | 39 | 33 | 238
  >= 65 years | 5 | 8 | 7 | 7 | 7 | 9 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 14 | 24 | 18 | 15 | 115
  Male | 30 | 34 | 41 | 31 | 37 | 40 | 213

OUTCOME MEASURES:

1. Primary Outcome: Baseline Hemoglobin A1c (HbA1c)
Description: HbA1c is measured as percent.
Time Frame: Baseline
Population: All randomized participants.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 54 | 54 | 55 | 55 | 55 | 55
Percent | 8.08 (0.14) | 8.01 (0.17) | 7.88 (0.13) | 8.13 (0.17) | 8.30 (0.16) | 8.24 (0.15)

2. Primary Outcome: Change From Baseline in HbA1c at Week 12
Description: HbA1c is measured as percent. The change from baseline is the Week 12 HbA1c percent minus the Week 0 HbA1c percent (last observation carried forward [LOCF]).
Time Frame: Baseline and Week 12
Population: Analysis population included randomized participants who were treated, had a baseline HbA1c measurement and at least 1 post-baseline HbA1c measurement up to Week 12.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 53
Percent | -0.11 [-0.25 to 0.04] | -0.56 [-0.69 to -0.42] | -0.80 [-0.94 to -0.66] | -0.73 [-0.87 to -0.58] | -0.83 [-0.98 to -0.69] | -0.87 [-1.01 to -0.73]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; The null hypothesis is that there is no difference between ertugliflozin and placebo on the primary endpoint; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.45, 80% CI 2-sided [-0.65 to -0.25]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; The null hypothesis is that there is no difference between ertugliflozin and placebo on the primary endpoint; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.69, 80% CI 2-sided [-0.89 to -0.49]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; The null hypothesis is that there is no difference between ertugliflozin and placebo on the primary endpoint; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.62, 80% CI 2-sided [-0.82 to -0.42]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; The null hypothesis is that there is no difference between ertugliflozin and placebo on the primary endpoint; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.72, 80% CI 2-sided [-0.93 to -0.52]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.76, 80% CI 2-sided [-0.97 to -0.56]

3. Secondary Outcome: Change From Baseline in HbA1C at Week 2
Description: HbA1c is measured as percent. The change from baseline is the Week 2 HbA1c percent minus the Week 0 HbA1c percent (LOCF).
Time Frame: Baseline and Week 2
Population: Analysis population included randomized participants who were treated, had a baseline HbA1c measurement and at least 1 post-baseline HbA1c measurement up to Week 2.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 52 | 49 | 50 | 49 | 51
Percent | 0.00 [-0.08 to 0.07] | -0.14 [-0.21 to -0.06] | -0.29 [-0.36 to -0.21] | -0.22 [-0.29 to -0.15] | -0.17 [-0.25 to -0.10] | -0.26 [-0.33 to -0.18]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.049, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.13, 80% CI 2-sided [-0.24 to -0.03]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.29, 80% CI 2-sided [-0.39 to -0.18]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.22, 80% CI 2-sided [-0.32 to -0.11]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.020, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.17, 80% CI 2-sided [-0.27 to -0.06]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.25, 80% CI 2-sided [-0.36 to -0.15]

4. Secondary Outcome: Change From Baseline in HbA1c at Week 4
Description: HbA1c is measured as percent. The change from baseline is the Week 4 HbA1c percent minus the Week 0 HbA1c percent (LOCF).
Time Frame: Baseline and Week 4
Population: Analysis population included randomized participants who were treated, had a baseline HbA1c measurement and at least 1 post-baseline HbA1c measurement up to Week 4.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 53
Percent | -0.04 [-0.13 to 0.06] | -0.40 [-0.50 to -0.31] | -0.49 [-0.59 to -0.40] | -0.48 [-0.57 to -0.38] | -0.40 [-0.49 to -0.30] | -0.48 [-0.57 to -0.38]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.37, 80% CI 2-sided [-0.50 to -0.23]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.45, 80% CI 2-sided [-0.59 to -0.32]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.44, 80% CI 2-sided [-0.57 to -0.30]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.36, 80% CI 2-sided [-0.49 to -0.22]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.44, 80% CI 2-sided [-0.57 to -0.30]

5. Secondary Outcome: Change From Baseline in HbA1c at Week 8
Description: HbA1c is measured as percent. The change from baseline is the Week 8 HbA1c percent minus the Week 0 HbA1c percent (LOCF).
Time Frame: Baseline and Week 8
Population: Analysis population included randomized participants who were treated, had a baseline HbA1c measurement and at least 1 post-baseline HbA1c measurement up to Week 8.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 53
Percent | -0.10 [-0.22 to -0.02] | -0.57 [-0.69 to -0.45] | -0.76 [-0.88 to -0.64] | -0.73 [-0.85 to -0.60] | -0.75 [-0.87 to -0.62] | -0.77 [-0.89 to -0.65]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.47, 80% CI 2-sided [-0.64 to -0.30]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.66, 80% CI 2-sided [-0.83 to -0.49]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.63, 80% CI 2-sided [-0.80 to -0.45]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.65, 80% CI 2-sided [-0.82 to -0.47]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.67, 80% CI 2-sided [-0.84 to -0.50]

6. Secondary Outcome: Baseline Body Weight
Time Frame: Baseline
Population: All randomized participants.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 54 | 54 | 55 | 55 | 55 | 55
kg | 83.78 (2.37) | 83.44 (2.57) | 85.74 (2.82) | 82.28 (2.93) | 81.81 (2.34) | 85.52 (2.61)

7. Secondary Outcome: Percent Change From Baseline in Body Weight at Week 12
Description: The percent change from baseline is the ([Week 12 body weight minus the Week 0 body weight] divided by the Week 0 body weight) X 100 (LOCF).
Time Frame: Baseline and Week 12
Population: Analysis population included randomized participants who were treated, had a baseline body weight measurement and at least 1 post-baseline body weight measurement up to Week 12.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent change
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 53
Percent change | -0.75 [-1.18 to -0.32] | -1.90 [-2.32 to -1.48] | -2.50 [-2.92 to -2.07] | -2.90 [-3.33 to -2.47] | -2.66 [-3.10 to -2.23] | -0.30 [-0.72 to 0.13]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.007, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.15, 80% CI 2-sided [-1.75 to -0.55]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.75, 80% CI 2-sided [-2.35 to -1.14]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.15, 80% CI 2-sided [-2.76 to -1.54]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.91, 80% CI 2-sided [-2.52 to -1.30]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.833, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = 0.45, 80% CI 2-sided [-0.15 to 1.06]

8. Secondary Outcome: Percent Change From Baseline in Body Weight at Week 2
Description: The percent change from baseline is the ([Week 2 body weight minus the Week 0 body weight] divided by the Week 0 body weight) X 100 (LOCF).
Time Frame: Baseline and Week 2
Population: Analysis population included randomized participants who were treated, had a baseline body weight measurement and at least 1 post-baseline body weight measurement up to Week 2.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent change
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 52 | 48 | 50 | 49 | 50
Percent change | -0.24 [-0.46 to -0.02] | -0.65 [-0.87 to -0.44] | -1.36 [-1.59 to -1.14] | -1.14 [-1.36 to -0.92] | -1.11 [-1.33 to -0.88] | 0.21 [-0.01 to 0.43]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.043, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.42, 80% CI 2-sided [-0.73 to -0.11]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.13, 80% CI 2-sided [-1.44 to -0.81]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.90, 80% CI 2-sided [-1.22 to -0.59]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.87, 80% CI 2-sided [-1.18 to -0.55]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.967, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = 0.45, 80% CI 2-sided [0.14 to 0.76]

9. Secondary Outcome: Percent Change From Baseline in Body Weight at Week 4
Description: The percent change from baseline is the ([Week 4 body weight minus the Week 0 body weight] divided by the Week 0 body weight) X 100 (LOCF).
Time Frame: Baseline and Week 4
Population: Analysis population included randomized participants who were treated, had a baseline body weight measurement and at least 1 post-baseline body weight measurement up to Week 4.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent change
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 52
Percent change | -0.44 [-0.73 to -0.15] | -1.20 [-1.48 to -0.92] | -1.76 [-2.04 to -1.48] | -1.68 [-1.97 to -1.39] | -1.52 [-1.81 to -1.23] | 0.01 [-0.28 to 0.30]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.008, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.76, 80% CI 2-sided [-1.17 to -0.36]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.32, 80% CI 2-sided [-1.73 to -0.91]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.24, 80% CI 2-sided [-1.65 to -0.83]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Odds Ratio (OR) = -1.08, 80% CI 2-sided [-1.49 to -0.67]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.922, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Odds Ratio (OR) = 0.45, 80% CI 2-sided [0.04 to 0.86]

10. Secondary Outcome: Percent Change From Baseline in Body Weight at Week 8
Description: The percent change from baseline is the ([Week 8 body weight minus the Week 0 body weight] divided by the Week 0 body weight) X 100 (LOCF).
Time Frame: Baseline and Week 8
Population: Analysis population included randomized participants who were treated, had a baseline body weight measurement and at least 1 post-baseline body weight measurement up to Week 8.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent change
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 53
Percent change | -0.62 [-0.96 to -0.28] | -1.65 [-1.98 to -1.32] | -2.18 [-2.52 to -1.85] | -2.30 [-2.64 to -1.96] | -2.40 [-2.74 to -2.06] | -0.38 [-0.71 to -0.05]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.03, 80% CI 2-sided [-1.51 to -0.56]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.57, 80% CI 2-sided [-2.04 to -1.09]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.68, 80% CI 2-sided [-2.16 to -1.21]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.78, 80% CI 2-sided [-2.26 to -1.30]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.741, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = 0.24, 80% CI 2-sided [-0.24 to 0.71]

11. Secondary Outcome: Baseline Systolic Blood Pressure
Description: Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed.
Time Frame: Baseline
Population: All randomized participants.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 54 | 54 | 55 | 55 | 55 | 55
mmHg | 126.7 (1.71) | 126.5 (2.18) | 127.9 (2.31) | 125.8 (1.97) | 124.9 (2.20) | 126.6 (1.83)

12. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 12
Description: Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed. The change from baseline is the Week 12 systolic blood pressure minus the Week 0 systolic blood pressure (LOCF).
Time Frame: Baseline and Week 12
Population: Analysis population included randomized participants who were treated, had a baseline systolic blood pressure measurement and at least 1 post-baseline systolic blood pressure measurement up to Week 12.
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 53
mmHg | -0.55 [-2.55 to 1.44] | -2.69 [-4.63 to -0.75] | -4.03 [-5.99 to -2.07] | -3.43 [-5.43 to -1.43] | -3.93 [-5.94 to -1.91] | -1.09 [-3.05 to 0.87]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.163, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.13, 80% CI 2-sided [-4.92 to 0.65]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.056, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -3.48, 80% CI 2-sided [-6.28 to -0.68]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.096, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.88, 80% CI 2-sided [-5.70 to -0.05]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.064, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -3.37, 80% CI 2-sided [-6.21 to -0.53]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.403, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.54, 80% CI 2-sided [-3.33 to 2.26]

13. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 2
Description: Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed. The change from baseline is the Week 2 systolic blood pressure minus the Week 0 systolic blood pressure (LOCF).
Time Frame: Baseline and Week 2
Population: Analysis population included randomized participants who were treated, had a baseline systolic blood pressure measurement and at least 1 post-baseline systolic blood pressure measurement up to Week 2.
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 52 | 49 | 50 | 49 | 50
mmHg | -1.93 [-3.73 to -0.12] | -2.30 [-4.08 to -0.51] | -4.73 [-6.57 to -2.89] | -2.28 [-4.10 to -0.45] | -5.39 [-7.23 to -3.55] | -0.91 [-2.74 to 0.91]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.425, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.37, 80% CI 2-sided [-2.91 to 2.17]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.082, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.81, 80% CI 2-sided [-5.38 to -0.23]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.430, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.35, 80% CI 2-sided [-2.92 to 2.21]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.043, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -3.47, 80% CI 2-sided [-6.05 to -0.89]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.694, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = 1.01, 80% CI 2-sided [-1.55 to 3.58]

14. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 4
Description: Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed. The change from baseline is the Week 4 systolic blood pressure minus the Week 0 systolic blood pressure (LOCF).
Time Frame: Baseline and Week 4
Population: Analysis population included randomized participants who were treated, had a baseline systolic blood pressure measurement and at least 1 post-baseline systolic blood pressure measurement up to Week 4.
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 52
mmHg | -2.57 [-4.31 to -0.82] | -3.94 [-5.64 to -2.25] | -5.15 [-6.86 to -3.44] | -5.43 [-7.17 to -3.69] | -3.33 [-5.09 to -1.57] | -3.32 [-5.05 to -1.60]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.234, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.38, 80% CI 2-sided [-3.81 to 1.05]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.087, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.59, 80% CI 2-sided [-5.03 to -0.14]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.068, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.86, 80% CI 2-sided [-5.33 to -0.40]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.346, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.77, 80% CI 2-sided [-3.25 to 1.71]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.346, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.76, 80% CI 2-sided [-3.21 to 1.70]

15. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 8
Description: Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed. The change from baseline is the Week 8 systolic blood pressure minus the Week 0 systolic blood pressure (LOCF).
Time Frame: Baseline and Week 8
Population: Analysis population included randomized participants who were treated, had a baseline systolic blood pressure measurement and at least 1 post-baseline systolic blood pressure measurement up to Week 8.
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 53
mmHg | -0.44 [-2.42 to 1.55] | -1.53 [-3.46 to 0.40] | -2.85 [-4.80 to -0.90] | -3.04 [-5.03 to -1.06] | -3.30 [-5.31 to -1.30] | -2.43 [-4.38 to -0.48]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.306, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.10, 80% CI 2-sided [-3.87 to 1.67]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.133, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.41, 80% CI 2-sided [-5.19 to 0.37]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.117, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.61, 80% CI 2-sided [-5.42 to 0.20]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.097, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.87, 80% CI 2-sided [-5.69 to -0.04]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.179, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.00, 80% CI 2-sided [-4.78 to 0.79]

16. Secondary Outcome: Baseline Diastolic Blood Pressure
Description: as for outcome 11
Time Frame: Baseline
Population: All randomized participants.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 54 | 54 | 55 | 55 | 55 | 55
mmHg | 79.14 (1.24) | 78.95 (1.14) | 78.19 (1.36) | 78.45 (1.32) | 78.61 (1.24) | 79.15 (1.01)

17. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 12
Description: Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed. The change from baseline is the Week 12 diastolic blood pressure minus the Week 0 diastolic blood pressure (LOCF).
Time Frame: Baseline and Week 12
Population: Analysis population included randomized participants who were treated, had a baseline diastolic blood pressure measurement and at least 1 post-baseline diastolic blood pressure measurement up to Week 12.
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 53
mmHg | 0.81 [-0.41 to 2.02] | -1.12 [-2.30 to 0.06] | -1.01 [-2.20 to 0.18] | -3.18 [-4.40 to -1.97] | -1.83 [-3.06 to -0.61] | 1.68 [0.49 to 2.87]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.072, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.93, 80% CI 2-sided [-3.62 to -0.24]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.086, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.81, 80% CI 2-sided [-3.51 to -0.11]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -3.99, 80% CI 2-sided [-5.71 to -2.27]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.025, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.64, 80% CI 2-sided [-4.37 to -0.92]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.746, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = 0.88, 80% CI 2-sided [-0.82 to 2.58]

18. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 2
Description: Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed. The change from baseline is the Week 2 diastolic blood pressure minus the Week 0 diastolic blood pressure (LOCF).
Time Frame: Baseline and Week 2
Population: Analysis population included randomized participants who were treated, had a baseline diastolic blood pressure measurement and at least 1 post-baseline diastolic blood pressure measurement up to Week 2.
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 52 | 49 | 50 | 49 | 50
mmHg | -0.57 [-1.69 to 0.56] | -1.25 [-2.37 to -0.14] | -1.26 [-2.41 to -0.12] | -1.97 [-3.11 to -0.84] | -3.01 [-4.16 to -1.86] | 0.92 [-0.22 to 2.06]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.289, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.69, 80% CI 2-sided [-2.27 to 0.90]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.288, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.70, 80% CI 2-sided [-2.31 to 0.91]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.130, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.41, 80% CI 2-sided [-3.01 to 0.19]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.026, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.44, 80% CI 2-sided [-4.05 to -0.84]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.883, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = 1.49, 80% CI 2-sided [-0.11 to 3.08]

19. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 4
Description: Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed. The change from baseline is the Week 4 diastolic blood pressure minus the Week 0 diastolic blood pressure (LOCF).
Time Frame: Baseline and Week 4
Population: Analysis population included randomized participants who were treated, had a baseline diastolic blood pressure measurement and at least 1 post-baseline diastolic blood pressure measurement up to Week 4.
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 52
mmHg | -0.80 [-1.80 to 0.21] | -2.47 [-3.44 to -1.49] | -3.08 [-4.07 to -2.10] | -2.81 [-3.81 to -1.80] | -2.10 [-3.11 to -1.09] | -0.51 [-1.51 to 0.48]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.063, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.67, 80% CI 2-sided [-3.07 to -0.27]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.019, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.29, 80% CI 2-sided [-3.69 to -0.88]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.035, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.01, 80% CI 2-sided [-3.43 to -0.59]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.121, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.30, 80% CI 2-sided [-2.73 to 0.12]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.602, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = 0.29, 80% CI 2-sided [-1.13 to 1.70]

20. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 8
Description: Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed. The change from baseline is the Week 8 diastolic blood pressure minus the Week 0 diastolic blood pressure (LOCF).
Time Frame: Baseline and Week 8
Population: Analysis population included randomized participants who were treated, had a baseline diastolic blood pressure measurement and at least 1 post-baseline diastolic blood pressure measurement up to Week 8.
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 53
mmHg | 0.80 [-0.40 to 1.99] | -1.40 [-2.56 to -0.24] | -0.69 [-1.86 to 0.48] | -2.23 [-3.42 to -1.04] | -1.20 [-2.40 to 0.01] | 0.32 [-0.85 to 1.49]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.045, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -2.20, 80% CI 2-sided [-3.86 to -0.54]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.126, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.49, 80% CI 2-sided [-3.16 to 0.18]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.011, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -3.03, 80% CI 2-sided [-4.72 to -1.34]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.066, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -1.99, 80% CI 2-sided [-3.69 to -0.30]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.357, ANCOVA — P-value is one-sided; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -0.48, 80% CI 2-sided [-2.15 to 1.19]

21. Secondary Outcome: Baseline Fasting Plasma Glucose
Description: Laboratory measurements were performed after an overnight fast ≥8 hours in duration.
Time Frame: Baseline
Population: All randomized participants.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 54 | 54 | 55 | 55 | 55 | 55
mg/dL | 165.3 (5.65) | 162.5 (6.75) | 156.5 (5.79) | 163.3 (6.30) | 171.3 (7.69) | 166.2 (6.70)

22. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 12
Description: The change from baseline is the Week 12 FPG minus the Week 0 fasting plasma glucose (LOCF). Laboratory measurements were performed after an overnight fast ≥8 hours in duration.
Time Frame: Baseline and Week 12
Population: Analysis population included randomized participants who were treated, had a baseline fasting plasma glucose measurement and at least 1 post-baseline fasting plasma glucose measurement up to Week 12.
Measure: Least Squares Mean (80% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 53
mg/dL | 2.76 [-2.47 to 8.00] | -18.23 [-23.32 to -13.14] | -23.06 [-28.21 to -17.90] | -31.47 [-36.71 to -26.24] | -29.26 [-34.58 to -23.94] | -17.29 [-22.43 to -12.15]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -20.99, 80% CI 2-sided [-28.29 to -13.69]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided.P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -25.82, 80% CI 2-sided [-33.17 to -18.47]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -34.23, 80% CI 2-sided [-41.64 to -26.83]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -32.02, 80% CI 2-sided [-39.49 to -24.56]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -20.05, 80% CI 2-sided [-27.39 to -12.72]

23. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 2
Description: The change from baseline is the Week 2 FPG minus the Week 0 FPG (LOCF). Laboratory measurements were performed after an overnight fast ≥8 hours in duration.
Time Frame: Baseline and Week 2
Population: Analysis population included randomized participants who were treated, had a baseline fasting plasma glucose measurement and at least 1 post-baseline fasting plasma glucose measurement up to Week 2.
Measure: Least Squares Mean (80% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 51 | 49 | 50 | 49 | 51
mg/dL | 5.89 [0.50 to 11.27] | -15.07 [-20.46 to -9.69] | -15.68 [-21.19 to -10.17] | -26.65 [-32.09 to -21.21] | -16.44 [-21.97 to -10.91] | -14.69 [-20.07 to -9.30]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -20.96, 80% CI 2-sided [-28.58 to -13.34]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -21.57, 80% CI 2-sided [-29.27 to -13.86]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -32.54, 80% CI 2-sided [-40.20 to -24.88]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -22.33, 80% CI 2-sided [-30.05 to -14.61]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -20.57, 80% CI 2-sided [-28.19 to -12.96]

24. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 4
Description: The change from baseline is the Week 4 FPG minus the Week 0 FPG (LOCF). Laboratory measurements were performed after an overnight fast ≥8 hours in duration.
Time Frame: Baseline and Week 4
Population: Analysis population included randomized participants who were treated, had a baseline fasting plasma glucose measurement and at least 1 post-baseline fasting plasma glucose measurement up to Week 4.
Measure: Least Squares Mean (80% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 53
mg/dL | 5.17 [0.10 to 10.24] | -16.91 [-21.84 to -11.99] | -22.77 [-27.77 to -17.78] | -27.95 [-33.02 to -22.88] | -26.62 [-31.77 to -21.46] | -18.00 [-22.98 to -13.03]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -22.09, 80% CI 2-sided [-29.16 to -15.01]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -27.94, 80% CI 2-sided [-35.06 to -20.83]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -33.12, 80% CI 2-sided [-40.29 to -25.95]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -31.79, 80% CI 2-sided [-39.02 to -24.56]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -23.17, 80% CI 2-sided [-30.28 to -16.07]

25. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 8
Description: The change from baseline is the Week 8 FPG minus the Week 0 FPG (LOCF). Laboratory measurements were performed after an overnight fast ≥8 hours in duration.
Time Frame: Baseline and Week 8
Population: Analysis population included randomized participants who were treated, had a baseline fasting plasma glucose measurement and at least 1 post-baseline fasting plasma glucose measurement up to Week 8.
Measure: Least Squares Mean (80% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 51 | 54 | 53 | 51 | 50 | 53
mg/dL | 3.82 [-1.06 to 8.69] | -18.25 [-22.99 to -13.51] | -24.69 [-29.49 to -19.89] | -31.59 [-36.46 to -26.71] | -30.99 [-35.94 to -26.04] | -18.93 [-23.71 to -14.15]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -22.07, 80% CI 2-sided [-28.87 to -15.27]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -28.51, 80% CI 2-sided [-35.35 to -21.67]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 10 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -35.40, 80% CI 2-sided [-42.30 to -28.51]
Statistical Analysis 4: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -34.81, 80% CI 2-sided [-41.76 to -27.86]
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value is rounded to 3 decimals; therefore, p <0.0005 is reported as 0.000; ANCOVA model with treatment as fixed effect and baseline as covariate with last observation carried forward; Difference in least squares means = -22.75, 80% CI 2-sided [-29.58 to -15.92]

26. Secondary Outcome: Percentage of Participants Achieving HbA1c <7% at Week 12
Description: Laboratory measurements were performed after an overnight fast ≥8 hours in duration.
Time Frame: Week 12
Population: Analysis population excludes participants with missing Week 12 HbA1c measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 45 | 50 | 49 | 44 | 47 | 51
Percentage of participants | 15.6 | 44.0 | 42.9 | 38.6 | 36.2 | 43.1

27. Secondary Outcome: Percentage of Participants Achieving HbA1C <6.5% at Week 12
Description: Laboratory measurements were performed after an overnight fast ≥8 hours in duration.
Time Frame: Week 12
Population: Analysis population excludes participants with missing Week 12 HbA1c measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 45 | 50 | 49 | 44 | 47 | 51
Percentage of participants | 6.7 | 12.0 | 20.4 | 13.6 | 14.9 | 25.5

28. Secondary Outcome: Number of Participants Who Experienced an Advere Event (AE)
Description: An adverse event is defines as any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. Below table includes all data collected since the first dose of sponsor-provided metformin.
Time Frame: Up to 98 days
Population: All participants who received at least 1 dose of treatment (including sponsor-supplied metformin).
Measure: Number; unit: Participants
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg | Metformin Run-in
Number analyzed (Participants) | 54 | 54 | 55 | 55 | 55 | 55 | 375
Participants | 29 | 31 | 30 | 29 | 28 | 30 | 82

29. Secondary Outcome: Number of Participants Who Discontinued Study Medication Due to an AE
Description: An adverse event is defines as any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. Below table includes all data collected since the first dose of sponsor-provided metformin and excludes a temporary discontinuation of study medication.
Time Frame: Up to 84 days
Population: All participants who received at least 1 dose of treatment (including sponsor-supplied metformin).
Measure: Number; unit: Participants
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg | Metformin Run-in
Number analyzed (Participants) | 54 | 54 | 55 | 55 | 55 | 55 | 375
Participants | 1 | 1 | 3 | 2 | 1 | 1 | 3

ADVERSE EVENTS:
Time Frame: Up to 24 weeks (including 10-week run-in period, 12-week treatment period, and 2-week follow-up period).
Description: Data presented below include the metformin run-in group (run-in period), 6 treatment groups (treatment period) and no upper limit on the follow-up window for participants who discontinued study drug.
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 10 mg | Ertugliflozin 25 mg | Sitagliptin 100 mg | Metformin Run-in
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54 | 2/55 | 0/55 | 1/55 | 1/55 | 2/375
Other Adverse Events (participants affected / at risk) | 13/54 | 10/54 | 14/55 | 14/55 | 10/55 | 12/55 | 30/375
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | Ertugliflozin 1 mg (N=54) | Ertugliflozin 5 mg (N=55) | Ertugliflozin 10 mg (N=55) | Ertugliflozin 25 mg (N=55) | Sitagliptin 100 mg (N=55) | Metformin Run-in (N=375)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | Ertugliflozin 1 mg (N=54) | Ertugliflozin 5 mg (N=55) | Ertugliflozin 10 mg (N=55) | Ertugliflozin 25 mg (N=55) | Sitagliptin 100 mg (N=55) | Metformin Run-in (N=375)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 14 (14)
Genital infection fungal (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 3 (4) | 4 (4) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 1 (2) | 4 (4)
Blood pressure increased (Investigations) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 6 (6) | 2 (2) | 2 (2) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator will provide manuscripts, abstracts, or the full text of any other intended disclosure (poster presentation, invited speaker or guest lecturer presentation, etc.) to the Sponsor at least 30-days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, Investigator agrees to delay the disclosure for a period not to exceed an additional 60 days.